CLINICAL TRIAL: NCT02736461
Title: Factors Associated With Postoperative Strabismus After Floor Fracture Repair
Status: Completed | Type: Observational
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Ke-Hung Chien, Ophthalmologist, Tri-Service General Hospital
Other Study IDs: 1-104-05-124
Record Dates: First submitted 2016-03-18; First posted 2016-04-13 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Orbital Fractures; Strabismus
Keywords: Orbital fractures; Strabismus; Predicting factors; orbital floor fractures
MeSH Terms: conditions — Orbital Fractures; Strabismus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Group 1- With strabismus: Study group with strabismus happening after floor fracture repair
  Interventions: Procedure: Floor repair surgery
- Group 2- Without strabismus: No strabismus happening after floor fracture repair
  Interventions: Procedure: Floor repair surgery

INTERVENTIONS:
Procedure: Floor repair surgery

SUMMARY:
In patients suffered from floor fractures, there are 21.9% complaining about diplopia before fracture repair surgery and 20.8% after operation. Even after 6 months, there still are 16.4% had similar conditions. Investigators are planned to find predicting factors to prevent such conditions from happening.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from floor fractures in Tri-Service General Hospital in past 10 years.

Exclusion Criteria:

* Prior ocular surgeries
* Multiple facial trauma or facial bone fractures

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients suffering from floor fractures in Tri-Service General Hospital in past 10 years.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2016-07; Primary Completion 2017-10-12 (Actual); Study Completion 2017-10-12 (Actual)

PRIMARY OUTCOMES:
Strabismus happening | 6 months after orbital floor fracture repair surgery
  Number of participants suffered from strabismus happening at 6 months after operation and their characteristics.

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan

REFERENCES:
- [Result] Bartoli D, Fadda MT, Battisti A, Cassoni A, Pagnoni M, Riccardi E, Sanzi M, Valentini V. Retrospective analysis of 301 patients with orbital floor fracture. J Craniomaxillofac Surg. 2015 Mar;43(2):244-7. doi: 10.1016/j.jcms.2014.11.015. Epub 2014 Nov 29. PMID 25547215